CLINICAL TRIAL: NCT01029067
Title: Metacognitive Training (MCT) Compared With Cognitive Remediation (CR) in Schizophrenia: a Randomized Controlled Study Over 4 Weeks
Brief Title: Metacognitive Training in Schizophrenia
Acronym: MCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCT
Record Dates: First submitted 2009-12-05; First posted 2009-12-09 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Delusions; Schizophrenia
Keywords: schizophrenia; delusion; paranoia; psychosis
MeSH Terms: conditions — Delusions; Schizophrenia; Paranoid Disorders; Psychotic Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Remediation (Active Comparator): Computerized cognitive remediation (CogPack training). A fixed series is administered, which covers a wide range of neuropsychological exercises involving memory, reasoning, selective attention and psychomotor speed. The difficulty level for each patient is adapted automatically depending on to the subject's performance on prior exercises. At the end of each session, the patient receives individual feedback on his or her performance. To match with group MCT, eight sessions are administered. Each session lasts approximately 45-60 minutes.
  Interventions: Behavioral: Cognitive Remediation
- Metacognitive Training (Experimental): The group metacognitive training program (MCT) is fully documented (Moritz, Woodward, & Metacognition Study Group, 2007; VanHam Campus Press) and can be obtained in more than 15 languages cost-free via the following link: www.uke.de/mkt. The group program is delivered to groups of 3-10 patients by trained psychologists addressing delusion-related metacognitive biases (e.g., jumping to conclusions). The eight modules are presented via a video projector using pdf-converted Power-Point slides. Each group session lasts approximately 45-60 minutes. Individualized MCT (MCT+) follows group sessions and accords to the general guidelines for cognitive-behavioral therapy. For each patient, 8 one-to-one sessions were carried in addition to one session relating to the medical history.
  Interventions: Behavioral: Metacognitive training

INTERVENTIONS:
Behavioral: Metacognitive training — Group (8 sessions) and individualized metacognitive training (9 sessions), delivered by psychologists versus cognitive remediation (8 sessions) delivered by either psychologists or psychology students at an advanced master level
  Arms: Metacognitive Training
Behavioral: Cognitive Remediation — Group (8 sessions) and individualized metacognitive training (9 sessions), delivered by psychologists versus cognitive remediation (8 sessions) delivered by either psychologists or psychology students at an advanced master level
  Arms: Cognitive Remediation

SUMMARY:
Over a period of 4 weeks, metacognitive training for schizophrenia patients (MCT), delivered both in a group and individually, is compared to cognitive remediation (CogPack training). Blind to treatment assignment, both groups are assessed before intervention and four weeks later with the Positive and Negative Symptoms Scale (PANSS), the Psychosis Rating Scales (PSYRATS) and cognitive tests. Delusion severity serves as the primary endpoint. It is assumed that MCT will improve delusion severity to a greater extent than CR in the course of 4 weeks taking medication into account.

DETAILED DESCRIPTION:
Metacognitive training for schizophrenia patients (MCT) is a manualized group intervention that can be obtained cost-free online. MCT seeks to sharpen the awareness of schizophrenia spectrum patients on cognitive biases (e.g. jumping to conclusions) contributing to delusion formation and maintenance and conveys cognitive strategies to counter these. The present trial combines group MCT with an individualized cognitive-behavioral oriented approach entitled MCT+. Patients with schizophrenia are randomly allocated to either metacognitive treatment (MCT) or cognitive remediation (CogPack training). Blind to treatment assignment, both groups are assessed prior to intervention and four weeks later with the Positive and Negative Symptoms Scale (PANSS), the Psychosis Rating Scales (PSYRATS) and cognitive tasks. Delusion scores derived from the PANSS and PSYRATS serve as main outcome parameters. We also explore if MCT improves jumping to conclusions with a probabilistic reasoning task. To make results as generalizable as possible to a typical inpatient population, broad inclusion criteria are chosen. Patients are only excluded if age is < 18 and > 65 years and diagnoses do not meet criteria of a schizophrenia spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia spectrum disorder

Exclusion Criteria:

* intellectual disability (IQ < 70)
* unable to provide informed consent
* hostility on PANSS > 4
* suspiciousness on PANSS > 5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
delusion severity as assessed with the Positive and Negative Syndrome Scale (PANSS); sum of item scores p1, p5, p6 and g9 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Moritz, PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg Eppendorf, Hamburg, Hamburg, Germany

REFERENCES:
- See also: link to metacognitive training site, where training material can be downloaded cost-free — http://www.uke.de/mkt